CLINICAL TRIAL: NCT06058312
Title: Evaluation of Changes in Adherence to the Mediterranean Diet in Cancer Patients Undergoing Treatment
Brief Title: Individual Food Preferences for the Mediterranean Diet in Cancer Patients
Acronym: MyPrefMed
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Antoine Lacassagne (Other)
Collaborators: University of Lyon (Other); University of Firenze and Siena, Napoli, Italy (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2022/34
Record Dates: First submitted 2023-08-21; First posted 2023-09-28 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Neoplasms
MeSH Terms: conditions — Neoplasms | interventions — Health

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental Arms (Experimental)
  Interventions: Other: Self-questionnaire

INTERVENTIONS:
Other: Self-questionnaire — The self-administered questionnaires to be completed at the time of inclusion will be presented to the patient on a tablet during the inclusion visit and will be completed on the same day in the Day Hospital using the Compusense software. Online self-questionnaires and sensory tests at the 9th week of treatment will also be conducted using the Compusense software in small groups at a designated location within the center.
  Other Names: sensory tests
Other: Self-questionnaire — The MediLite questionnaire consists of nine items that assess daily consumption of fruits, vegetables, grains, meats and meat products, dairy products, alcohol, and olive oil, as well as weekly consumption of legumes and fish.
  Other Names: MediLite adhérence score
Other: Self-questionnaire — The CITAS is a self-administered questionnaire consisting of 18 items evaluated on a five-point Likert scale and divided into three dimensions: 1) quantitative changes in taste perception (hypogeusia and ageusia), 2) qualitative changes in taste perception (heterogeusia, cacogeusia), and 3) nutrition-related problems (difficulty eating hot or fatty foods).
  Using a Likert scale ranging from 1 to 5 (where 1 = no difficulty or absence of disturbance and 5 = maximum difficulty or disturbance), CITAS assesses the four dimensions of taste disturbances: taste intensity, discomfort, phantogeusia, and parageusia, as well as overall taste alterations.
  For the original version by Kano and Kanda (2013), five items assessing changes in smell from the modified CITAS version by Drareni et al. 2021 will be added in this study.
  Other Names: Chemotherapy-induced Taste Alterations CITAS
Other: Self-questionnaire — Food neophobia will be assessed using the Food Neophobia Scale (FNS) developed by Pliner & Hobden (1992). The FNS consists of ten statements evaluated on a 7-point agreement scale ranging from 1 = "I strongly disagree" to 7 = "I strongly agree." Individual FNS scores are calculated as the sum of the ratings given to the ten statements after reversing the neophilic items; thus, scores theoretically range from 10 to 70, with higher scores reflecting higher levels of food neophobia.
  Other Names: FNS -Food Neophobia scale
Other: Self-questionnaire — The quality of life related to food in cancer patients is composed of 46 items with a 4-point scale (never, almost never, almost always, always). The questionnaire is divided into different subdomains: Cooking, where one eats and conviviality, Eating and drinking, After eating.
  Other Names: Food-Related Quality of Life in Cancer Patients
Other: Self-questionnaire — Individual baseline disgust sensitivity is assessed using the Disgust Sensitivity-Short Form (DS-SF) questionnaire; this questionnaire is a shortened version of the disgust scale aimed at measuring disgust of animal origin, based on contamination and revulsion (Haidt, 2004; Haidt et al., 1994; Inbar, Pizarro, and Bloom, 2009; Olatunji et al., 2007). This measure consists of 8 items divided into 2 parts. In the first part, statements were rated on a scale from 1 (not at all agree-very false about me) to 5 (completely agree-very true about me); for the second part, additional statements were rated from 1 (not at all disgusting) to 5 (extremely disgusting). The total disgust sensitivity score is obtained by summing the scores after two items have been reversed and ranges from 8 to 40.
  Other Names: Sensitivity to disgust
Other: Self-questionnaire — The subscale of reward sensitivity from the short version of reward and punishment sensitivity has been selected (17 items). Each item will be assessed on a 4-point Likert scale, ranging from 1 (completely no) to 4 (completely yes).
  Other Names: Short version Sensitivity to Reward Questionnaire
Other: Self-questionnaire — The EmoPrefMed questionnaire was developed to measure declared appreciation and emotional responses to selected Mediterranean diet (RM) products and changes in appreciation before and after chemotherapy.
  The assessment of the acceptability of a series of RM foods (listed in the questionnaire appendix) will be evaluated using a nine-point hedonic scale ranging from a minimum of 1 = "I don't like it at all" to a maximum of 9 = "I like it a lot" (Peryam & Pilgrim, 1957).
  Emotions will be assessed using a check-all-that-apply (CATA) list of emotions, including 4 negative and 4 positive emotions with low, moderate, and high arousal levels (It brings me joy, It intrigues me, It relaxes me, It annoys me, It leaves me indifferent, It makes me sad, It's monotonous, It disgusts me). Patients will be asked to select all the emotions they deem appropriate to describe the food product.
  Other Names: Questionnaire EmoPrefMed (Stated liking questionnaire et emotional profiling of selected MD products)
Other: Self-questionnaire — Food-related attitudes will be measured using the HTAS (Health and Taste Attitude Scale) proposed by Roininen et al. (1999), consisting of six subscales focusing on perceived health and taste aspects of foods. The two scales selected in this study are general interest in health (eight items, measuring overall interest in a healthy diet) and the use of food as a reward (six items, measuring attitudes towards using food as a reward). Each subscale consists of an equal number of statements phrased positively and negatively (Roininen et al., 1999). All items were rated on a seven-point category scale, ranging from "strongly disagree" to "strongly agree." As suggested by Roininen et al. (1999), negative statements were reversed and recoded for the calculation of final scores.
  Other Names: Health and taste attitude scale
Other: Self-questionnaire — The response to PROP (6-n-propyl-2-thiouracil) is measured using 1.5 cm diameter paper disks previously soaked in a solution of deionized water with a concentration of 3.2 mM PROP, dissolving 0.5477 g/L of PROP. Each paper disk will contain approximately 0.280 mg of PROP. Participants are asked to place the paper disk on the tip of their tongue for 20 seconds, then remove it and assess the perceived bitter intensity on a Labelled Magnitude Scale (LMS).
  The LMS scale consists of a vertical line of 100 units with labels placed at no sensation, 0; barely detectable, 1.4; weak, 6; moderate, 17; strong, 34.7; very strong, 52.5; and the strongest imaginable sensation of any kind, 100. Numeric labels are not reported on the scale. Participants are instructed to think of the "strongest imaginable sensation" as the most intense sensation they can imagine in the realm of taste. Participants are encouraged to ask questions about the use of the scale if they need more clarification.
  Other Names: Taste test
Other: Self-questionnaire — The odors (Mint, Anise, Banana, Pine, Garlic, Cinnamon, Lemon) are trapped in tightly packed microcapsules (aminoplast type, diameter: 4-8 μm). Microcapsule-based ink is printed on cardboard paper (SILK-250 g; Size: 11 cm × 21 cm). Each odorant has been printed in a defined area (2 cm in diameter). The odor is released by simply rubbing the printed microcapsule reserve (scratch-and-sniff method).Patients receive a disposable single-use sample and are asked to identify the odors and evaluate on a visual analog scale the perceived intensity, perceived irritation, and appreciation of each odor.
  Other Names: Olfactory Test
Other: Self-questionnaire — Two model foods were developed to investigate responses to variations in sweetness, acidity, and freshness. The first range consists of Apple-Mint Juice, composed of four samples containing different concentrations of mint syrup (0, 15, 60, 240 g/kg). The second range is a chickpea mousse made up of four samples containing different quantities of citric acid and glucose-fructose syrup (glucose-fructose syrup: 0, 50, 100, 200 g/kg; citric acid: 8, 6, 4, 4 g/kg). Participants are asked to evaluate the samples using the Labelled Affective Magnitude Scale. Regarding the LAM scale, subjects are instructed to consider the extremes of appreciation, "the best I can imagine" and "the worst I can imagine". After a break, they are asked to taste the samples again and rate the intensity of sweetness, acidity, apple flavor, mint flavor, and freshness on the Labeled Magnitude Scale: from 'not detectable' to 'the strongest imaginable'.
  Other Names: Test for the Evaluation of Food Products from the Mediterranean Diet

SUMMARY:
This is an exploratory study aimed at characterizing adherence to the Mediterranean diet among patients undergoing treatment for cancer, in relation to sensory alterations that occur during treatment.

The primary strength of this project lies in the consideration of a large number of variables that scientific literature has shown to play a significant role in the dietary behavior of patients. The project's multidisciplinary approach, which takes into account both sensory perception and psychological dimensions, can enrich scientific knowledge on the subject, enabling a better understanding of the dietary behaviors of cancer patients undergoing treatment.

One of the main strengths of the project is that taste and smell reactivity will be tested using a combined approach that includes the evaluation of responses to PROP (Propylthiouracil - a bitter compound), selected aromas and odors, responses to model foods belonging to the Mediterranean diet in which the intensities of selected sensory properties are expected to be affected by chemotherapy (e.g., sweetness and freshness).

To date, no study has investigated adherence to the Mediterranean diet in such a wide range of patients. The choice of a Mediterranean diet framework is based on evidence defining this type of diet as a health promoter, improving health and preventing diseases and health complications. The Mediterranean diet includes the food variety present in the specific region chosen for the study, ensuring variety and availability of local products. The selection of the Antoine Lacassagne Center in Nice is based on the need to study the dietary preferences of a Mediterranean population familiar with Mediterranean diet products.

This project could serve as the foundation for a dietary development aspect, in which foods adapted to cancer patients will be created and tested to mitigate issues of malnutrition.

Expected Benefits Addressing the scientific question regarding the impact of sensory and psychological variables on adherence to the Mediterranean Diet and dietary behavior of cancer patients undergoing treatment will help identify individual variables to consider in assisting patients in adopting health-promoting behavior and reducing malnutrition.

Expected Risks The research project does not involve maneuvers or the implementation of care procedures other than those to which patients would be subjected if they were not participating in the study. This research involves no specific risks, except for possible risks of allergies or food intolerances related to the sensory testing session. The dietary models used only include food ingredients normally available in markets.

In order to test the taste sensitivity index, the response to propylthiouracil (PROP) will be evaluated using paper discs previously soaked in a solution composed of water and PROP according to the method of Zhao et al. (2003). This procedure has been safely used in children as well as in several studies (including patients undergoing chemotherapy) approved by ethics committees in multiple institutes from various countries.

Scientific Impact The project will provide information about the variables that impact the dietary behavior of patients undergoing chemotherapy. This knowledge will be useful in developing principles that contribute to reducing malnutrition rates in oncology patients.

Methodology This is an exploratory study aimed at characterizing adherence to the Mediterranean diet among patients with cancer undergoing treatment, who may experience changes in their relationship with food as well as their dietary behavior. Adherence to the Mediterranean diet will be studied in cancer patients at T0 (before the start of treatment) and at T1 (after 9 weeks of treatment). A comparison will be made between patients without sensory alterations and patients with taste and/or smell alterations at T1. The psychological and sensory variables impacting dietary behavior will also be measured and correlated with adherence to the Mediterranean diet and the presence or absence of sensory alterations.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged 18-70 years old,
* Patient cared for at the Center Antoine Lacassagne (CAL) Day Hospital and needing to start chemotherapy or immunotherapy,
* Patient to return to the Antoine Lacassagne center in their 9th week of therapy,
* Patient who has not received chemotherapy or specific treatment in the 3 months prior to inclusion (wash-out period of 3 months),
* Patient having read the information note and having attested to his non-objection
* Patient not having objected to the use of this data in the context of medical research
* Patient affiliated with a Social Security scheme.

Exclusion Criteria:

* Inability to eat, or patient with enteral/parenteral nutrition,
* Patient who has undergone gastric surgery,
* Patient undergoing radiotherapy at the level of the ENT sphere (due to the possibility of affection of the mouth due to the RTH),
* Patient with cancer of the ENT sphere (upper aerodigestive tract),
* Patient with an allergy or intolerance to one of the foods offered during the sensory test sessions
* Vulnerable persons as defined in article L1121-5 to -8:
* Pregnant women, parturients and breastfeeding mothers,
* Persons deprived of their liberty by a judicial or administrative decision, persons hospitalized without consent under Articles L. 3212-1 and L. 3213-1 who do not fall under the provisions of Article L. 1121-8,
* and persons admitted to a health or social establishment for purposes other than research,
* Adults subject to a legal protection measure or unable to express their consent.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 442 (Estimated)
Dates: Start 2023-09-04 (Actual); Primary Completion 2024-09-04 (Estimated); Study Completion 2024-09-04 (Estimated)

PRIMARY OUTCOMES:
role of sensory alterations | 9 weeks
  The primary outcome measure of the study is the reduction in adherence score to the Mediterranean diet between T0, at inclusion, and T1, after 9 ± 2 weeks of treatment. The difference in the reduction of scores between T0 and T1 will be compared for two groups of subjects (to be formed at T1): those who report sensory alterations and those who do not. The total score of sensory alterations will be calculated based on the CiTAS questionnaire - Chemotherapy-induced Taste Alterations (Kano & Kanda, 2013). A threshold of 1.5 will be used to distinguish patients reporting taste or smell alterations (≥1.5) from those not reporting them (<1.5), following Di Meglio et al. (2022).
  The analysis will be conducted by comparing the MediLite score before and after 9 weeks of treatment for patients with or without sensory alterations (threshold 1.5 CITAS score).

SECONDARY OUTCOMES:
Taste perception | 9 weeks
  Investigate the taste perception (response to PROP, a bitter compound). The individual scores of response to PROP (propylthiouracil, a bitter compound) using the LMS (Labelled Magnitude Scale)
olfactory perception | 9 weeks
  Investigate the olfactory perception (Sniff & scratch of 7 smells). The individual scores of response to odors using the Olfactory Test.
Liking for Mediterranean-type | 9 weeks
  Explore the relationship between liking for Mediterranean-type products . The individual food appreciation scores (four variants of hummus and four variants of apple-mint juice) using the LAM (Labelled Affective Magnitude Scale).
Perceived intensity of sensations for Mediterranean-type | 9 weeks
  The individual scores for the perception of the intensity of food sensations (four variants of hummus and four variants of apple-mint juice) using the LMS (Labelled Magnitude Scale).
Food neophobia | 9 weeks
  Investigate food neophobia (FNS) with "Food Neophobia Scale (FNS) in cancer patients undergoing treatment.
Dietary Quality of life | 9 weeks
  Investigate dietary quality of life (QVA score) in cancer patients undergoing treatment
relationships to health and food attitude | 9 weeks
  Investigate relationships to health (general health interest-HTAS) and food (food as a reward-HTAS)
Sensitivity to Reward | 9 weeks
  Investigate Sensitivity to Reward (SPSRQ)
Sensitivity to disgust | 9 weeks
  Investigate Sensitivity to Disgust (DS-SF)
Liking and emotions mediterranean food | 9 weeks
  Investigate food liking (9 hedonic point scale) and emotion (CATA emotions) using tje EmoPrefMEd questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Antoine lacassagne, Nice, France

IPD SHARING:
Plan to Share IPD: Undecided